CLINICAL TRIAL: NCT04780919
Title: The Ultrasound-Monitored Changes in Achilles Tendinopathy After Focused Extracorporeal Shock Wave Therapy - a Randomized Sham-Controlled Trial
Brief Title: Ultrasound-Monitored Changes in Achilles Tendinopathy After Extracorporeal Shock Wave Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Stanislav Machač, Ph.D, Academic worker, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK- 1/21
Record Dates: First submitted 2021-02-24; First posted 2021-03-04 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Achilles Tendinopathy
Keywords: Extracorporeal Shock Wave Therapy; Achilles Tendinopathy; Ultrasonography

STUDY DESIGN:
Intervention Model Description: Participants are divided into two groups - treatment and placebo.
Who Masked: Participant
Masking Description: Participants don't know which group (either treatment or placebo) they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (A) (Experimental): Group of patients with Achilles tendinopathy which are treated by focused extracorporeal shockwave therapy once a week for 5 weeks. ESWT parameters: 0,12 mJ/mm2, 10 Hz, 1300 shocks.
  Interventions: Device: BTL-6000 FSWT
- Sham Group (B) (Sham Comparator): Group of patients with Achilles tendinopathy in which sham extracorporeal shockwave therapy is applied once a week for 5 weeks. Total applications are 5, applicated weekly. Sham ESWT parameters are same as in Group A (0,12 mJ/mm2, 10 Hz, 1300 shocks) but with modified applicator which does not allow wave transmission.
  Interventions: Device: BTL-6000 FSWT with sham applicator

INTERVENTIONS:
Device: BTL-6000 FSWT — Intensity 0,12 mJ/mm2, frequency 10 Hz, total number of shocks 1300.
  Arms: Treatment Group (A)
Device: BTL-6000 FSWT with sham applicator — Intensity 0,12 mJ/mm2, frequency 10 Hz, total number of shocks 1300 - applied with modified applicator which does not allow wave transmission.
  Arms: Sham Group (B)

SUMMARY:
This study is designed as a randomized, placebo-controlled clinical trial in which we monitor the effects of low-energy focused extracorporeal shockwave therapy (ESWT) in patients with Achilles tendinopathy (AT). Participants will be randomly divided into two groups. ESWT according to selected parameters will be applied to Group A. Group B will receive sham ESWT.

Patients in both groups will have the same program. The research for one patient lasts a total of 8 weeks (2 months) from the initial to the final examination. In the first week, there will be a clinical examination by a physiotherapist, an ultrasonographic examination, and the patient will complete a VISA-A questionnaire. At the end of the examination, the patient will be randomly assigned to group A or B and receive the first application. For the next 4 weeks, additional applications will be performed once a week. The interval between individual applications should be at least 7 days. Thus, a total of 5 applications of ESWT or sham ESWT will be performed. The final examination will take place 3 weeks after the last application and will include the same procedures as for the initial examination.

DETAILED DESCRIPTION:
This study is designed as a randomized, placebo-controlled clinical trial in which we monitor the effects of low-energy focused extracorporeal shockwave therapy (ESWT) in patients with Achilles tendinopathy (AT). Participants will be randomly divided into two groups. ESWT according to selected parameters will be applied to Group A. Group B will receive sham ESWT.

Patients in both groups will have the same program. The research for one patient lasts a total of 8 weeks (2 months) from the initial to the final examination. In the initial session, there will be a clinical examination by a physiotherapist, which includes case history questions, measuring range of motion (measured by weight-bearing lunge test), functional loading tests (1-leg heel rise test, 1-leg hop test) and an ultrasonographic examination (tendon cross section area and width at the maximal tendon antero-posterior width place). In addition, the patient will complete a VISA-A questionnaire. At the end of the initial session, the patient will be randomly assigned to group A or B and receive the first application. For the next 4 weeks, additional applications will be performed once a week. The interval between individual applications should be at least 7 days. Thus, a total of 5 applications of ESWT or sham ESWT will be performed. The final examination will take place 3 weeks after the last application and will include the same procedures as for the initial examination.

ELIGIBILITY:
Inclusion Criteria:

* the patient complains about Achilles tendon pain, which limits (at least partially) his quality of life during daily activities or sport, and this condition would be referred as a tendinopathy
* the patient's other leg is asymptomatic
* the patient is not aware of the symptomatical mechanical tendon damage in past (eg. partial or complete rupture due to injury)
* the patient has no previous experience with extracorporeal shockwave therapy treatment

Exclusion Criteria:

* the patient has condition which is contraindication for extracorporeal shock wave therapy treatment
* the patient had symptomatical mechanical tendon damage in past (eg. partial or complete rupture due to injury)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Machač, Mgr., Ph.D., Principal Investigator — University Hospital Motol and 2nd Faculty of Medicine, Charles University
Locations (1):
- University Hospital Motol and 2nd Faculty of Medicine, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group (A): Group of assigned patients with Achilles tendinopathy which were treated by focused extracorporeal shockwave therapy once a week for 5 weeks.
  BTL-6000 FSWT: Intensity 0,12 mJ/mm2, frequency 10 Hz, total number of shocks 1300.
- Sham Group (B): Group of assigned patients with Achilles tendinopathy in which sham extracorporeal shockwave therapy is applied once a week for 5 weeks. Total applications are 5, applicated weekly. Sham ESWT parameters are same as in Group A (0,12 mJ/mm2, 10 Hz, 1300 shocks) but with modified applicator which does not allow wave transmission.
  BTL-6000 FSWT with sham applicator: Intensity 0,12 mJ/mm2, frequency 10 Hz, total number of shocks 1300 - applied with modified applicator which does not allow wave transmission.
Period: Overall Study
Arm/Group | Treatment Group (A) | Sham Group (B)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group (A) | Sham Group (B) | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (9.6) | 43.2 (12.3) | 39.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (4.4) | 32.7 (7.5) | 29.6 (6.8)
Duration of difficulties [Mean (Standard Deviation); unit: months] — Simple question about duration of experienced difficulties until the baseline assessment. The result answer is presented in whole number of months. A number equal to 12 months refers the duration of the difficulties equal to or longer than 1 year.
  months | 6 (3.8) | 7.6 (4.4) | 6.8 (4.1)
Baseline maximal pain [Mean (Standard Deviation); unit: units on a scale] — Using Numeric Rating Scale in points reaching 0-10. Higher points indicate worse pain.
  units on a scale | 6.6 (1.7) | 6.1 (2.3) | 6.3 (2)
Baseline VISA-A score [Mean (Standard Deviation); unit: score on a scale] — Using the Victorian Institute of Sports Assessment - Achilles questionaire. Higher score indicates better condition.
  score on a scale | 64.3 (12.1) | 65.3 (15.9) | 64.8 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cross-sectional Area at the Place of Maximum Tendon Width
Description: Measured by measuring tools in ultrasound machine in cm2. In linear view is selected maximal width place, then the position of ultrasound head is rotated to horizontal view and in this view cross section area is measured.
Time Frame: Change of initial values at 3 weeks follow up after last application (8th week).
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Treatment Group (A) | Sham Group (B)
Number analyzed (Participants) | 9 | 9
cm^2
  Baseline | 0.8 (0.19) | 0.76 (0.18)
  3 weeks follow up after last application | 0.78 (0.2) | 0.69 (0.14)
Statistical Analysis 1: Comparison: Treatment Group (A) vs Sham Group (B); The Group A will have significantly decreased Cross Section Area compared to Group B at 3 weeks follow up after last application; Test type: Superiority; p = 0.722, Two-way ANOVA — p-value is adjusted to comparison between the Group A and Group B at 3 weeks follow-up after the last application

2. Primary Outcome: Change in Maximum Pain in the Achilles Tendon Area
Description: Measured by numeric rating scale in points. The values can reach 0-10 points. A higher score means worse pain.
Time Frame: Change in maximum pain in the timeframe of the last application (5th week)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group (A) | Sham Group (B)
Number analyzed (Participants) | 9 | 9
units on a scale
  Baseline | 6.6 (1.7) | 6.1 (2.3)
  Timeframe of last application | 3.6 (1.4) | 5.2 (1.9)
Statistical Analysis 1: Comparison: Treatment Group (A) vs Sham Group (B); The maximum pain will decrease significantly more in Group A compared to Group B in the timeframe of the last application compared to baseline; Test type: Superiority; p = 0.096, Two-way ANOVA — p-value is adjusted to comparison between the Group A and Group B in the timeframe of the last application

3. Primary Outcome: Change in Maximum Pain in the Achilles Tendon Area (Follow up)
Description: Measured by numeric rating scale in points. The values can reach 0-10 points. A higher score means worse pain.
Time Frame: Change in maximum pain at 3 weeks follow up after last application (8th week).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group (A) | Sham Group (B)
Number analyzed (Participants) | 9 | 9
units on a scale
  Baseline | 6.6 (1.7) | 6.1 (2.3)
  3 weeks follow up after last application | 2.7 (1.8) | 5 (2.1)
Statistical Analysis 1: Comparison: Treatment Group (A) vs Sham Group (B); The maximum pain will decrease significantly more in Group A compared to Group B at the 3 weeks follow up compared to baseline; Test type: Superiority; p = 0.035, Two-way ANOVA — p-value is adjusted to comparison between the Group A and Group B at the 3 weeks follow up compared to baseline

4. Primary Outcome: Change of Ankle Dorsiflexion Range of Motion
Description: Measured using weight-bearing lunge test in cm.
Time Frame: Change of initial values at 3 weeks follow up after last application (8th week).
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Treatment Group (A) | Sham Group (B)
Number analyzed (Participants) | 9 | 9
cm
  Baseline | 7.4 (3) | 8.7 (2.9)
  3 weeks follow up after last application | 10.1 (2.5) | 8.7 (3)
Statistical Analysis 1: Comparison: Treatment Group (A) vs Sham Group (B); The maximum of ankle dorsiflexion range of motion will increase significantly more in Group A compared to Group B at the 3 weeks follow up compared to baseline; Test type: Superiority; p = 0.171, Two-way ANOVA — p-value is adjusted to comparison between the Group A and Group B at the 3 weeks follow up compared to baseline

5. Secondary Outcome: Number of Participants With Hypoechogenic Areas
Description: Echostructure is evaluated visually by investigator using musculoskeletal ultrasound machine. Patients who have a hypoechogenic areas in the tendon are counted.
Time Frame: Change of the echostructure at 3 weeks follow up after last application (8th week).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group (A) | Sham Group (B)
Number analyzed (Participants) | 9 | 9
Participants
  Baseline | 6 | 6
  3 weeks follow up after last application | 6 | 6

6. Secondary Outcome: Number of Participants With Increased Thickness of Achilles Tendon
Description: The Achilles tendon continuity in evaluated visually by investigator using musculoskeletal ultrasound machine. Patients who have a visually significant increased thickness of tendon will be counted.
Time Frame: Change of the tendon continuity at 3 weeks follow up after last application (8th week).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group (A) | Sham Group (B)
Number analyzed (Participants) | 9 | 9
Participants
  Baseline | 5 | 4
  3 weeks follow up after last application | 5 | 4

7. Secondary Outcome: Change in VISA-A Questionnaire Score
Description: The VISA-A questionnaire is standardized questionnaire for patients with Achilles tendinopathy. The results are recorded in points (0-100 points). The higher score indicates patients better condition.
Time Frame: Change of initial values at 3 weeks follow up after last application (8th week).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group (A) | Sham Group (B)
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 64.3 (12.1) | 65.3 (15.9)
  3 weeks follow up after last application | 84.9 (9.9) | 69.2 (20)
Statistical Analysis 1: Comparison: Treatment Group (A) vs Sham Group (B); The VISA-A score will increase significantly more in Group A compared to Group B at the 3 weeks follow up compared to baseline; Test type: Superiority; p = 0.104, Two-way ANOVA — p-value is adjusted to comparison between the Group A and Group B in 3 weeks follow up after the last application

8. Secondary Outcome: Change in Single Leg Heel Rise Test
Description: Patient performs as many heel rises using only one leg as possible in 30 seconds or until first sign of pain in Achilles tendon area.
Time Frame: Change of initial values at 3 weeks follow up after last application (8th week)
Population: In the Group A, this test was performed by all participants in initial and final examination. In the Group B, this test was performed by all participants in initial examination and by 8 (of 9) participants in final examination. One patient was not able to perform this test in final examination due to the associated health complications (not caused by the used intervention).
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | Treatment Group (A) | Sham Group (B)
Number analyzed (Participants) | 9 | 8
repetitions
  Baseline | 16.6 (5.8) | 21.8 (10.8)
  3 weeks follow up after last application | 26.4 (7.6) | 26.5 (17.4)

9. Secondary Outcome: Change in Single Leg Hop Test
Description: Patient performs as many hops on one leg as possible in 30 seconds or until first sign of pain in Achilles tendon area.
Time Frame: Change of initial values at 3 weeks follow up after last application (8th week).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | Treatment Group (A) | Sham Group (B)
Number analyzed (Participants) | 9 | 8
repetitions
  Baseline | 31.1 (16.9) | 29.5 (23.6)
  3 weeks follow up after last application | 51.9 (12.7) | 45.0 (23.5)

ADVERSE EVENTS:
Time Frame: From baseline to 3 weeks follow up
Description: All-Cause Mortality is not expected when applying the ESWT at Achilles tendon area and was not monitored/assessed. However, Serious, and Other (Not Including Serious) Adverse Events were monitored using simple questions to patients during and after the procedure.
Arm/Group | Treatment Group (A) | Sham Group (B)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT04780919/Prot_SAP_000.pdf